CLINICAL TRIAL: NCT05301322
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF RESPIRATORY SYNCYTIAL VIRUS PREFUSION F SUBUNIT VACCINE WHEN COADMINISTERED WITH SEASONAL INACTIVATED INFLUENZA VACCINE IN ADULTS ≥65 YEARS OF AGE
Brief Title: Safety and Immunogenicity of RSVpreF Coadministered With SIIV in Adults ≥65 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3671006
Record Dates: First submitted 2022-03-02; First posted 2022-03-29 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Respiratory Syncytial Virus
Keywords: Respiratory tract infection; RSV; vaccine; older adults
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blinded.
  The participant, study coordinator, and all site staff will be blinded.
  The majority of sponsor staff will be blinded to study intervention allocation. All laboratory testing personnel performing serological assays or diagnostic assays will remain blinded to the study intervention assigned/received throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Coadministration Group (Experimental): RSVpreF and SIIV followed by placebo a month later
  Interventions: Biological: RSVpreF Vaccine; Other: Placebo; Biological: Seasonal Inactivated Influenza Vaccine
- Sequential Administration Group (Experimental): Placebo and SIIV followed by RSVpreF a month later
  Interventions: Biological: RSVpreF Vaccine; Other: Placebo; Biological: Seasonal Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: RSVpreF Vaccine — RSV Vaccine
Other: Placebo — Placebo
Biological: Seasonal Inactivated Influenza Vaccine — SIIV

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of RSVpreF when coadministered with SIIV compared to sequential administration of the vaccines when given 1 month apart (SIIV followed by RSVpreF). Additionally, the study will contribute data supporting the development of RSVpreF as a prophylactic vaccine against RSV disease in infants through maternal immunization and in older adults through active vaccination.

DETAILED DESCRIPTION:
This Phase 3, multicenter, parallel-group, placebo-controlled, randomized, double-blind study will be conducted in Australia and/or another southern hemisphere country.

Healthy adults ≥65 years of age will be randomized 1:1 to either the coadministration group (RSVpreF + SIIV)/placebo or the sequential-administration group (placebo + SIIV)/RSVpreF. This study design intends to use a single lot of NIP SIIV that is specifically indicated for use in adults ≥65 years of age.

There are 3 scheduled study visits each 1 month apart. To assess immunogenicity, 30 mL blood will be collected prior to vaccination at Visit 1 and Visit 2, and at Visit 3.

Local reactions (redness, swelling, and pain at the injection site) occurring at the RSVpreF or placebo injection site (left deltoid) and systemic events (fever, headache, fatigue, nausea, vomiting, diarrhea, muscle pain, and joint pain) occurring within 7 days after each vaccination visit (Visit 1 and Visit 2) will be prompted for and collected daily by the participant in an e-diary device or smartphone app. SIIV injection site reactions will not be routinely collected in the e-diary.

AEs and SAEs will be collected from the signing of informed consent through Visit 3.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥65 years of age at the time of consent.
2. Participants who are willing and able to comply with scheduled visits, laboratory tests, lifestyle considerations, and other study procedures, including daily completion of the e diary for 7 days after each study vaccination.
3. Healthy participants who are determined by medical history, physical examination and clinical judgment of the investigator to be eligible for inclusion in the study.
4. Capable of giving signed informed consent

Exclusion Criteria:

1. Bleeding diathesis or condition associated with prolonged bleeding time that may contraindicate IM injection.
2. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention or any related vaccine.
3. Allergy to egg proteins (egg or egg products) or chicken proteins.
4. History of Guillain-Barré syndrome.
5. Serious chronic disorder, including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
6. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
7. Other medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior, or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Previous vaccination with any licensed or investigational RSV vaccine at any time prior to enrollment, or planned receipt throughout the study of nonstudy RSV vaccine.
9. Previous vaccination with any influenza vaccine within 6 months before study intervention administration, or planned receipt of any nonstudy licensed or investigational influenza vaccine during study participation.
10. Receipt of any blood/plasma products or immunoglobulin, from 60 days before study intervention administration, or planned receipt throughout the study.
11. Individuals who receive chronic treatment with immunosuppressive therapy, including cytotoxic agents, monoclonal antibodies, systemic corticosteroids, or radiotherapy, eg, for cancer or an autoimmune disease, from 60 days before study intervention administration or planned receipt throughout the study. If systemic corticosteroids (<20 mg/day of prednisone or equivalent) have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled in the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intra articular, intrabursal, or topical (skin or eyes) corticosteroid use is permitted.
12. Current alcohol abuse or illicit drug use.
13. Current use of any prohibited concomitant medication(s) or those unwilling/unable to use a permitted concomitant medication(s)
14. Participation in other studies involving investigational product(s) within 28 days prior to consent and/or during study participation
15. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1471 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- Australia (33):
  - Paratus Clinical Research Canberra, Bruce, Australian Capital Territory
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Emeritus Research, Botany, New South Wales
  - Genesis Research Services, Broadmeadow, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Northside Health, Coffs Harbour, New South Wales
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - The AIM Centre / Hunter Diabetes Centre, Merewether, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Scientia Clinical Research, Randwick, New South Wales
  - Australian Clinical Research Network, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Paratus Clinical Research Brisbane, Albion, Queensland
  - Core Research Group, Brisbane, Queensland
  - Griffith University, Gold Coast Campus, Queensland
  - Nucleus Network Brisbane, Herston, Queensland
  - Mackay Hospital and Health Service, Mackay, Queensland
  - USC Clinical Trials Moreton Bay, Morayfield, Queensland
  - USC Clinical Trials Centre, Sippy Downs, Queensland
  - AusTrials - Taringa, Taringa, Queensland
  - Core Research Group, Taringa, Queensland
  - AusTrials Wellers Hill, Tarragindi, Queensland
  - CMAX Clinical Research Pty Ltd, Adelaide, South Australia
  - University of Tasmania, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Emeritus Research, Camberwell, Victoria
  - Barwon Health, Geelong, Victoria
  - Doctors of Ivanhoe, Ivanhoe, Victoria
  - Nucleus Network Brisbane, Melbourne, Victoria
  - Nucleus Network Melbourne, Melbourne, Victoria
  - Institute for Respiratory Health, Nedlands, Western Australia
  - Latitude Clinical Research, Spearwood, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Athan E, Baber J, Quan K, Scott RJ, Jaques A, Jiang Q, Li W, Cooper D, Cutler MW, Kalinina EV, Anderson AS, Swanson KA, Gruber WC, Gurtman A, Schmoele-Thoma B; Study C3671006 Investigator Group. Safety and Immunogenicity of Bivalent RSVpreF Vaccine Coadministered With Seasonal Inactivated Influenza Vaccine in Older Adults. Clin Infect Dis. 2024 May 15;78(5):1360-1368. doi: 10.1093/cid/ciad707. PMID 37992000
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671006

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1471 participants signed the informed consent and were enrolled in the study, of which 68 were screen failures and 1403 participants were randomized to a vaccine group.
Groups:
- (RSVpreF + SIIV)/Placebo: Coadministration Group: Participants were randomized to receive a single dose of seasonal inactivated influenza vaccine (SIIV) intramuscularly into the right deltoid muscle along with 120 micrograms (mcg) respiratory syncytial virus stabilized prefusion F subunit vaccine (RSVpreF) intramuscularly into the left deltoid muscle (Vaccination 1) on Day 1; and placebo intramuscularly into the left deltoid muscle (Vaccination 2) after 1 month. Participants were followed up for 1 month after Vaccination 2.
- (Placebo + SIIV)/RSVpreF: Sequential-Administration Group: Participants were randomized to receive a single dose of SIIV intramuscularly into the right deltoid muscle along with placebo intramuscularly into the left deltoid muscle (Vaccination 1) on Day 1; and 120 mcg RSVpreF intramuscularly into the left deltoid muscle (Vaccination 2) after 1 month. Participants were followed up for 1 month after Vaccination 2.
Period: Overall Study
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Started | 705 | 698 (1 participant received SIIV but was discontinued prior to receiving placebo at Vaccination 1 (as randomized) and is thus not included in the safety tables.)
Not Vaccinated | 3 (Participants were counted as not completed study due to the following reasons: protocol violation (2 participants) and other unspecified (1 participant).) | 1 (Participant was counted as not completed study due to protocol violation.)
Vaccination 1 | 702 | 697
Vaccination 2 | 688 | 693
Completed | 686 | 692
Not Completed | 19 | 6
Not completed — Adverse Event | 7 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Other | 4 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received the study intervention (RSVpreF, placebo, or SIIV). The safety population was based on study intervention actually received. One participant randomized in the Sequential-Administration Group incorrectly received RSVpreF + SIIV at Vaccination 1; hence, the participant was included in the vaccine group as administered i.e., (RSVpreF + SIIV)/Placebo: Coadministration Group.
Groups:
- Total: Total of all reporting groups
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group | Total
Number analyzed (Participants) | 703 | 696 | 1399
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.7 (4.7) | 70.7 (4.7) | 70.7 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 398 | 372 | 770
  Male | 305 | 324 | 629
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 652 | 647 | 1299
  Unknown or Not Reported | 46 | 41 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 22 | 21 | 43
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 7
  Black or African American | 0 | 0 | 0
  White | 669 | 665 | 1334
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Vaccination With RSVpreF or Placebo
Description: Local reactions were collected at the RSVpreF or placebo injection site after Vaccination 1 and Vaccination 2 and were recorded by participants using electronic diary (e-diary). Local reactions included redness, swelling and pain at injection site. Redness and swelling were measured and recorded in measuring device units where, 1 measuring device unit =0.5 centimeter (cm) and were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), and severe (>10.0 cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity). Percentage of participants reporting local reactions at injection site in Coadministration Group, and Sequential-Administration Group and associated 2-sided 95% confidence interval (CI) based on Clopper and Pearson method was presented in this outcome measure (OM). Safety population=all enrolled participants who received study intervention (RSVpreF, placebo).
Time Frame: Within 7 days after Vaccination 1 or Vaccination 2
Population: Safety population was analyzed. 'Overall Number of Participants (Par) Analyzed' (N)= par with at least 1 e-diary (within 7 days through Vaccination [vax]) transmitted. 1 par randomized in Sequential-Administration Group (SAG) incorrectly received RSVpreF + SIIV at Vax 1; hence, par was included in (RSVpreF + SIIV)/Placebo. 1 par randomized in SAG incorrectly received placebo at Vax 2; hence, par was included in vaccine group administered at Vax 1 and excluded from safety analysis at Vax 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RSVpreF + SIIV: Coadministration Group: On Day 1 (Visit 1), participants received a single dose of seasonal inactivated influenza vaccine (SIIV) intramuscularly into the right deltoid muscle along with 120 micrograms (mcg) respiratory syncytial virus stabilized prefusion F subunit vaccine (RSVpreF) intramuscularly into the left deltoid muscle (Vaccination 1).
- Placebo: Coadministration Group: One month after Vaccination 1, participants received placebo intramuscularly into the left deltoid muscle (Vaccination 2).
- Placebo + SIIV: Sequential-Administration Group: On Day 1 (Visit 1), participants received a single dose of SIIV intramuscularly into the right deltoid muscle along with placebo intramuscularly into the left deltoid muscle (Vaccination 1).
- RSVpreF: Sequential-Administration Group: One month after Vaccination 1, participants received 120 mcg RSVpreF intramuscularly into the left deltoid muscle (Vaccination 2).
Arm/Group | RSVpreF + SIIV: Coadministration Group | Placebo: Coadministration Group | Placebo + SIIV: Sequential-Administration Group | RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 701 | 681 | 693 | 686
Percentage of participants
  Pain at injection site: Mild | 10.1 [8.0 to 12.6] | 6.5 [4.7 to 8.6] | 7.6 [5.8 to 9.9] | 11.5 [9.2 to 14.1]
  Pain at injection site: Moderate | 1.3 [0.6 to 2.4] | 0.9 [0.3 to 1.9] | 0.7 [0.2 to 1.7] | 0.9 [0.3 to 1.9]
  Pain at injection site: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Redness: Mild | 2.1 [1.2 to 3.5] | 0.3 [0.0 to 1.1] | 0.6 [0.2 to 1.5] | 0.7 [0.2 to 1.7]
  Redness: Moderate | 0.9 [0.3 to 1.9] | 0.1 [0.0 to 0.8] | 0.1 [0.0 to 0.8] | 0.9 [0.3 to 1.9]
  Redness: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Swelling: Mild | 1.6 [0.8 to 2.8] | 0.3 [0.0 to 1.1] | 0.1 [0.0 to 0.8] | 1.2 [0.5 to 2.3]
  Swelling: Moderate | 1.3 [0.6 to 2.4] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0.6 [0.2 to 1.5]
  Swelling: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0.1 [0.0 to 0.8]

2. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days After Vaccination With RSVpreF or Placebo
Description: Systemic events included fever, fatigue, headache, nausea, vomiting, diarrhea, muscle pain and joint pain and were recorded by participants using an e-diary. Fever was defined as an oral temperature >=38.0 degree Celsius (deg C) and categorized as >=38.0 to 38.4 deg C (mild), >38.4 to 38.9 deg C (moderate), >38.9 to 40.0 deg C (severe) and >40.0 deg C (grade 4). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily routine activity). Vomiting was graded mild: 1 to 2 times in 24 hours (h), moderate: >2 times in 24h, and severe: required intravenous hydration. Diarrhea was graded mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. Percentage of participants with systemic events within 7 days after each vaccination and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Within 7 days after Vaccination 1 or Vaccination 2
Population: Safety population= all enrolled participants who received study intervention (RSVpreF, placebo). N= participant with at least 1 e-diary (within 7 days through vax) transmitted. 1 participant randomized in SAG incorrectly received RSVpreF + SIIV at Vax 1; hence, participant was included in (RSVpreF + SIIV)/Placebo. 1 participant randomized in SAG incorrectly received placebo at Vax 2; hence,participant was included in vaccine group administered at Vax 1 and excluded from safety analysis at Vax 2.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | RSVpreF + SIIV: Coadministration Group | Placebo: Coadministration Group | Placebo + SIIV: Sequential-Administration Group | RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 701 | 681 | 693 | 686
Percentage of Participants
  Fever: Mild | 1.1 [0.5 to 2.2] | 0.7 [0.2 to 1.7] | 0.9 [0.3 to 1.9] | 1.0 [0.4 to 2.1]
  Fever: Moderate | 0.3 [0.0 to 1.0] | 0.1 [0.0 to 0.8] | 0.3 [0.0 to 1.0] | 0.1 [0.0 to 0.8]
  Fever: Severe | 0.4 [0.1 to 1.2] | 0 [0.0 to 0.5] | 0.3 [0.0 to 1.0] | 0 [0.0 to 0.5]
  Fever: Grade 4 (>40.0 deg C) | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Fatigue: Mild | 15.4 [12.8 to 18.3] | 10.1 [8.0 to 12.6] | 15.6 [13.0 to 18.5] | 11.5 [9.2 to 14.1]
  Fatigue: Moderate | 13.7 [11.2 to 16.5] | 7.5 [5.6 to 9.7] | 11.3 [9.0 to 13.8] | 7.0 [5.2 to 9.2]
  Fatigue: Severe | 0.9 [0.3 to 1.9] | 0 [0.0 to 0.5] | 0.3 [0.0 to 1.0] | 0.6 [0.2 to 1.5]
  Headache: Mild | 13.7 [11.2 to 16.5] | 10.4 [8.2 to 13.0] | 14.3 [11.8 to 17.1] | 10.6 [8.4 to 13.2]
  Headache: Moderate | 5.8 [4.2 to 7.9] | 4.6 [3.1 to 6.4] | 6.1 [4.4 to 8.1] | 5.4 [3.8 to 7.4]
  Headache: Severe | 0.1 [0.0 to 0.8] | 0.1 [0.0 to 0.8] | 0.6 [0.2 to 1.5] | 0.1 [0.0 to 0.8]
  Vomiting: Mild | 0.4 [0.1 to 1.2] | 0.3 [0.0 to 1.1] | 0.4 [0.1 to 1.3] | 1.0 [0.4 to 2.1]
  Vomiting: Moderate | 0.6 [0.2 to 1.5] | 0.1 [0.0 to 0.8] | 0.1 [0.0 to 0.8] | 0.1 [0.0 to 0.8]
  Vomiting: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Nausea: Mild | 4.4 [3.0 to 6.2] | 3.7 [2.4 to 5.4] | 4.6 [3.2 to 6.5] | 4.2 [2.8 to 6.0]
  Nausea: Moderate | 2.7 [1.6 to 4.2] | 1.0 [0.4 to 2.1] | 1.2 [0.5 to 2.3] | 1.2 [0.5 to 2.3]
  Nausea: Severe | 0.4 [0.1 to 1.2] | 0 [0.0 to 0.5] | 0.3 [0.0 to 1.0] | 0 [0.0 to 0.5]
  Diarrhea: Mild | 6.1 [4.5 to 8.2] | 3.2 [2.0 to 4.9] | 4.9 [3.4 to 6.8] | 4.5 [3.1 to 6.4]
  Diarrhea: Moderate | 2.0 [1.1 to 3.3] | 1.5 [0.7 to 2.7] | 1.2 [0.5 to 2.3] | 1.5 [0.7 to 2.7]
  Diarrhea: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0.1 [0.0 to 0.8] | 0.3 [0.0 to 1.0]
  Muscle pain: Mild | 10.1 [8.0 to 12.6] | 6.9 [5.1 to 9.1] | 7.5 [5.7 to 9.7] | 5.8 [4.2 to 7.9]
  Muscle pain: Moderate | 5.6 [4.0 to 7.5] | 2.1 [1.1 to 3.4] | 4.8 [3.3 to 6.6] | 3.5 [2.3 to 5.2]
  Muscle pain: Severe | 0.1 [0.0 to 0.8] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0.1 [0.0 to 0.8]
  Joint pain: Mild | 6.8 [5.1 to 9.0] | 5.1 [3.6 to 7.1] | 5.8 [4.2 to 7.8] | 4.2 [2.8 to 6.0]
  Joint pain: Moderate | 4.3 [2.9 to 6.1] | 2.2 [1.2 to 3.6] | 3.5 [2.2 to 5.1] | 2.8 [1.7 to 4.3]
  Joint pain: Severe | 0.4 [0.1 to 1.2] | 0 [0.0 to 0.5] | 0 [0.0 to 0.5] | 0.1 [0.0 to 0.8]

3. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) Within 1 Month After Vaccination 1
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs within 1 month after Vaccination 1 were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Within 1 month after Vaccination 1
Population: Safety population = all enrolled participants who received study intervention (RSVpreF, placebo). N = participants evaluable for this outcome measure. 1 participant randomized in SAG incorrectly received RSVpreF + SIIV at Vax 1; hence, participant was included in (RSVpreF + SIIV)/Placebo. 1 participant randomized in SAG incorrectly received placebo at Vax 2; hence, participant was included in vaccine group administered at Vax 1 and excluded from safety analysis at Vax 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 703 | 695
Percentage of participants | 21.9 [18.9 to 25.1] | 19.3 [16.4 to 22.4]

4. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) Within 1 Month After Vaccination 2
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs within 1 month after Vaccination 2 were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Within 1 month after Vaccination 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 689 | 691
Percentage of participants | 17.0 [14.3 to 20.0] | 16.6 [13.9 to 19.6]

5. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs) Within 1 Month After Vaccination 1
Description: An SAE was defined as an AE that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or nonpathogenic or that was considered to be an important medical event. Percentage of participants with SAEs and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented. Percentage of participants reporting SAEs within 1 month after Vaccination 1 were reported in this outcome measure.
Time Frame: Within 1 month after Vaccination 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 703 | 695
Percentage of participants | 1.1 [0.5 to 2.2] | 0.9 [0.3 to 1.9]

6. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs) Within 1 Month After Vaccination 2
Description: An SAE was defined as an AE that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or nonpathogenic or that was considered to be an important medical event. Percentage of participants with SAEs and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented. Percentage of participants reporting SAEs within 1 month after Vaccination 2 were reported in this outcome measure.
Time Frame: Within 1 month after Vaccination 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 689 | 691
Percentage of participants | 0.3 [0.0 to 1.0] | 0.7 [0.2 to 1.7]

7. Primary Outcome: Geometric Mean Ratio (GMR) of Neutralizing Titer (NTs) at 1 Month After Vaccination With RSVpreF for RSV Subfamily A and B in RSVpreF + SIIV Compared to RSVpreF Alone
Description: Geometric mean titer (GMT) of RSV A and RSV B neutralizing titers for the Coadministration Group and Sequential-Administration Group were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CI were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the lower limit of quantification (LLOQ) were set to 0.5*LLOQ. Geometric mean ratio (GMR) was reported in the statistical analysis section and was calculated as ratio of GMTs in the Coadministration Group to the Sequential-Administration Group.
Time Frame: 1 month after Vaccination 1 for Coadministration Group and 1 month after Vaccination 2 for Sequential-Administration Group
Population: Evaluable RSV immunogenicity population: eligible par who received study interventions (RSVpreF, placebo, or SIIV) as randomized at both Visit (V) 1 & V 2; had 1-month RSVpreF postvaccination (PV) blood collection 25-49 days after RSVpreF Vax; no major protocol violation from randomization through 1-month RSVpreF PV blood draw; had at least 1 valid & determinate assay result 1 month after RSVpreF Vax. N= par evaluable for this OM & 'Number Analyzed'(n) = par evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 681 | 671
Titer
  RSV A | 19709.9 [18445.0 to 21061.7] | 22817.1 [21284.8 to 24459.7]
  RSV B: number analyzed (Participants) | 680 | 670
  RSV B | 18384.5 [17093.1 to 19773.5] | 21621.4 [20071.6 to 23290.8]
Statistical Analysis 1: Comparison: (RSVpreF + SIIV)/Placebo: Coadministration Group vs (Placebo + SIIV)/RSVpreF: Sequential-Administration Group; RSV A; Test type: Non-Inferiority — Noninferiority was declared if the lower limit of the 2-sided 95% CI for the GMR (Coadministration Group to Sequential-Administration Group) was greater than 0.667 for both RSV A and RSV B NTs; GMR = 0.86, 95% CI 2-sided [0.785 to 0.951] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Coadministration minus Sequential-Administration) and the corresponding CIs (based on Student's t distribution)
Statistical Analysis 2: Comparison: (RSVpreF + SIIV)/Placebo: Coadministration Group vs (Placebo + SIIV)/RSVpreF: Sequential-Administration Group; RSV B; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; GMR = 0.85, 95% CI 2-sided [0.766 to 0.943] — [estimate comment as in outcome 7, analysis 1]

8. Primary Outcome: GMR of the Strain-Specific Hemagglutination Inhibition (HAI) Titers 1 Month After Vaccination With SIIV in the Coadministration Group to the Corresponding HAI Titers in the Sequential-Administration Group
Description: GMTs of strain-specific HAI titers for the Coadministration Group and Sequential-Administration Group were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. GMR was reported in the statistical analysis section and was calculated as ratio of GMT in the Coadministration Group to the Sequential-Administration Group.
Time Frame: 1 month after Vaccination 1
Population: Evaluable SIIV immunogenicity population: eligible participants who received study interventions (RSVpreF, placebo, or SIIV) as randomized with SIIV at Visit 1; had 1-month postvaccination blood collection 25-49 days after SIIV vaccination; no major protocol violation from randomization through 1-month postvaccination blood draw; had at least 1 valid and determinate assay result 1 month after SIIV vaccination. N= participants evaluable for this OM & n= participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 680 | 687
Titer
  HAI: H1N1 A/Victoria | 139.6 [128.8 to 151.2] | 162.2 [149.9 to 175.6]
  HAI: H3N2 A/Darwin: number analyzed (Participants) | 679 | 687
  HAI: H3N2 A/Darwin | 104.7 [96.3 to 113.8] | 136.4 [125.0 to 148.8]
  HAI: B/Austria: number analyzed (Participants) | 674 | 686
  HAI: B/Austria | 113.3 [103.2 to 124.3] | 126.3 [115.6 to 138.0]
  HAI: B/Phuket: number analyzed (Participants) | 679 | 687
  HAI: B/Phuket | 106.7 [98.7 to 115.4] | 123.2 [114.6 to 132.4]
Statistical Analysis 1: Comparison: (RSVpreF + SIIV)/Placebo: Coadministration Group vs (Placebo + SIIV)/RSVpreF: Sequential-Administration Group; HAI: H1N1 A/Victoria; Test type: Non-Inferiority — Noninferiority was declared if the lower limit of the 2-sided 95% CI for the GMR (Coadministration Group to Sequential-Administration Group) was greater than 0.667 for each of the 4 influenza strains; GMR = 0.86, 95% CI 2-sided [0.769 to 0.963] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: (RSVpreF + SIIV)/Placebo: Coadministration Group vs (Placebo + SIIV)/RSVpreF: Sequential-Administration Group; HAI: H3N2 A/Darwin; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; GMR = 0.77, 95% CI 2-sided [0.680 to 0.866] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: (RSVpreF + SIIV)/Placebo: Coadministration Group vs (Placebo + SIIV)/RSVpreF: Sequential-Administration Group; HAI: B/Austria; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; GMR = 0.90, 95% CI 2-sided [0.789 to 1.019] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: (RSVpreF + SIIV)/Placebo: Coadministration Group vs (Placebo + SIIV)/RSVpreF: Sequential-Administration Group; HAI: B/Phuket; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; GMR = 0.87, 95% CI 2-sided [0.779 to 0.964] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Geometric Mean of the Neutralizing Titers for RSV A and RSV B Before Vaccination and at 1 Month and 2 Months After Vaccination With RSVpreF
Description: GMT of neutralizing titers of RSV A and RSV B before vaccination, at 1 month and 2 months after vaccination was reported in this outcome measure. Assay results below the LLOQ were set to 0.5*LLOQ. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). For Sequential-Administration Group, the time point for 2 months after vaccination was not reported since the participants received RSVpreF at Vaccination 2 and were followed up for 1 month after Vaccination 2.
Time Frame: Coadministration Group: before RSVpreF vaccination, and 1 and 2 months after RSVpreF vaccination; Sequential-Administration Group: before RSVpreF vaccination (most recent serology results before RSVpreF) and 1 month after RSVpreF vaccination
Population: Evaluable RSV immunogenicity population: eligible participants who received study interventions (RSVpreF, placebo, or SIIV) as randomized at both V 1 & V 2; had 1-month RSVpreF PV blood collection 25-49 days after RSVpreF Vax; no major protocol violation from randomization through 1-month RSVpreF PV blood draw; had at least 1 valid and determinate assay result 1 month after RSVpreF Vax. 'N' = participants evaluable for this outcome measure and 'n' = participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 681 | 671
Titer
  RSV A: Before RSVpreF vaccination: number analyzed (Participants) | 681 | 670
  RSV A: Before RSVpreF vaccination | 1951.2 [1829.4 to 2081.2] | 1999.1 [1862.4 to 2145.8]
  RSV A: 1 Month after RSVpreF vaccination | 19709.9 [18445.0 to 21061.7] | 22817.1 [21284.8 to 24459.7]
  RSV A: 2 Months after RSVpreF vaccination: number analyzed (Participants) | 678 | 0
  RSV A: 2 Months after RSVpreF vaccination | 15357.5 [14395.8 to 16383.5] |
  RSV B: Before RSVpreF vaccination | 1810.2 [1695.7 to 1932.4] | 1807.6 [1683.0 to 1941.4]
  RSV B: 1 Month after RSVpreF vaccination: number analyzed (Participants) | 680 | 670
  RSV B: 1 Month after RSVpreF vaccination | 18384.5 [17093.1 to 19773.5] | 21621.4 [20071.6 to 23290.8]
  RSV B: 2 Months after RSVpreF vaccination: number analyzed (Participants) | 678 | 0
  RSV B: 2 Months after RSVpreF vaccination | 13681.7 [12749.1 to 14682.5] |

10. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of the NTs for RSV A and RSV B Before Vaccination and at 1 Month and 2 Months After Vaccination With RSVpreF
Description: GMFR of neutralizing titers of RSV A and RSV B before vaccination and at 1 month and 2 months after vaccination was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the Student's t distribution).
Time Frame: Coadministration Group: before RSVpreF vaccination, and 1 and 2 months after vaccination; Sequential-Administration Group: before RSVpreF vaccination (most recent serology results before RSVpreF) and 1 month after vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 681 | 670
Fold rise
  RSV A: 1 month after RSVpreF vaccination | 10.0 [9.28 to 10.87] | 11.4 [10.46 to 12.36]
  RSV A: 2 months after RSVpreF vaccination: number analyzed (Participants) | 678 | 0
  RSV A: 2 months after RSVpreF vaccination | 7.8 [7.27 to 8.42] |
  RSV B: 1 month after RSVpreF vaccination: number analyzed (Participants) | 680 | 670
  RSV B: 1 month after RSVpreF vaccination | 10.1 [9.38 to 10.97] | 12.0 [11.02 to 12.98]
  RSV B: 2 months after RSVpreF vaccination: number analyzed (Participants) | 678 | 0
  RSV B: 2 months after RSVpreF vaccination | 7.6 [7.03 to 8.12] |

11. Secondary Outcome: HAI Geometric Mean Titer (GMT) Before Vaccination and 1 Month After Vaccination With SIIV
Description: HAI GMT before vaccination and 1 month after vaccination with SIIV was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: Before SIIV vaccination, and 1 month after vaccination
Population: Evaluable SIIV immunogenicity population: eligible participants who received study interventions (RSVpreF, placebo, or SIIV) as randomized with SIIV at Visit 1; had 1-month PV blood collection 25-49 days after SIIV vaccination; no major protocol violation from randomization through 1-month PV blood draw; had at least 1 valid and determinate assay result 1 month after SIIV vaccination. 'N' = participants evaluable for this outcome measure and 'n' = participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 680 | 687
Titer
  H1N1 A/Victoria: Before SIIV Vaccination: number analyzed (Participants) | 678 | 684
  H1N1 A/Victoria: Before SIIV Vaccination | 48.8 [44.3 to 53.9] | 43.3 [39.2 to 47.8]
  H1N1 A/Victoria: 1 Month After SIIV Vaccination | 139.6 [128.8 to 151.2] | 162.2 [149.9 to 175.6]
  H3N2 A/Darwin: Before SIIV Vaccination: number analyzed (Participants) | 678 | 682
  H3N2 A/Darwin: Before SIIV Vaccination | 21.9 [20.2 to 23.7] | 21.7 [20.0 to 23.5]
  H3N2 A/Darwin: 1 Month After SIIV Vaccination: number analyzed (Participants) | 679 | 687
  H3N2 A/Darwin: 1 Month After SIIV Vaccination | 104.7 [96.3 to 113.8] | 136.4 [125.0 to 148.8]
  B/Austria: Before SIIV Vaccination: number analyzed (Participants) | 677 | 679
  B/Austria: Before SIIV Vaccination | 32.4 [29.3 to 35.8] | 31.0 [28.2 to 34.1]
  B/Austria: 1 Month After SIIV Vaccination: number analyzed (Participants) | 674 | 686
  B/Austria: 1 Month After SIIV Vaccination | 113.3 [103.2 to 124.3] | 126.3 [115.6 to 138.0]
  B/Phuket: Before SIIV Vaccination: number analyzed (Participants) | 680 | 683
  B/Phuket: Before SIIV Vaccination | 47.5 [43.3 to 52.0] | 49.7 [45.4 to 54.3]
  B/Phuket: 1 Month After SIIV Vaccination: number analyzed (Participants) | 679 | 687
  B/Phuket: 1 Month After SIIV Vaccination | 106.7 [98.7 to 115.4] | 123.2 [114.6 to 132.4]

12. Secondary Outcome: GMFR of Strain-Specific HAI Titers Before Vaccination and 1 Month After Vaccination With SIIV
Description: GMFR of strain-specific HAI titers before vaccination and 1 month after vaccination with SIIV was reported in this outcome measure. GMFRs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of fold rises (later time point over earlier time point) and the corresponding CIs (based on Student's t distribution).
Time Frame: Before SIIV vaccination, and 1 month after vaccination
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | (RSVpreF + SIIV)/Placebo: Coadministration Group | (Placebo + SIIV)/RSVpreF: Sequential-Administration Group
Number analyzed (Participants) | 679 | 684
Fold rise
  H1N1 A/Victoria: number analyzed (Participants) | 678 | 684
  H1N1 A/Victoria | 2.6 [2.37 to 2.85] | 3.3 [3.00 to 3.65]
  H3N2 A/Darwin: number analyzed (Participants) | 678 | 682
  H3N2 A/Darwin | 4.1 [3.78 to 4.49] | 5.4 [4.92 to 5.84]
  B/Austria: number analyzed (Participants) | 673 | 679
  B/Austria | 3.1 [2.80 to 3.32] | 3.5 [3.26 to 3.87]
  B/Phuket: number analyzed (Participants) | 679 | 683
  B/Phuket | 2.1 [1.95 to 2.23] | 2.3 [2.15 to 2.48]

ADVERSE EVENTS:
Time Frame: Local reactions (at the RSVpreF or placebo injection site) and systemic events (systematic assessment): Within 7 days after each vaccination. SAEs and other AEs: up to 1 month after Vaccination 1 and 2
Description: Same event may appear as non-SAE & SAE but are distinct events. Event may be serious in 1 par & non-serious in another or 1 par may have experienced both serious & non-serious events.Safety population was analyzed. 1 par randomized in SAG incorrectly received RSVpreF+SIIV at Vax 1;hence, par was included in (RSVpreF + SIIV)/Placebo.1 par randomized in SAG incorrectly received placebo at Vax 2; hence,par was included in vaccine group administered at Vax 1 & excluded from safety analysis at Vax 2.
Arm/Group | RSVpreF + SIIV: Coadministration Group | Placebo: Coadministration Group | Placebo + SIIV: Sequential-Administration Group | RSVpreF: Sequential-Administration Group
All-Cause Mortality (participants affected / at risk) | 0/703 | 0/689 | 1/695 | 0/691
Serious Adverse Events (participants affected / at risk) | 8/703 | 2/689 | 6/695 | 5/691
Other Adverse Events (participants affected / at risk) | 418/703 | 300/689 | 370/695 | 330/691
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSVpreF + SIIV: Coadministration Group (N=703) | Placebo: Coadministration Group (N=689) | Placebo + SIIV: Sequential-Administration Group (N=695) | RSVpreF: Sequential-Administration Group (N=691)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Amaurosis fugax (Eye disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSVpreF + SIIV: Coadministration Group (N=703) | Placebo: Coadministration Group (N=689) | Placebo + SIIV: Sequential-Administration Group (N=695) | RSVpreF: Sequential-Administration Group (N=691)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Episcleritis (Eye disorders) | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Macular oedema (Eye disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1
Fatigue (FATIGUE) (General disorders) | 210 | 120 | 188 | 131
Feeling hot (General disorders) | 0 | 0 | 2 | 0
Influenza like illness (General disorders) | 1 | 3 | 3 | 1
Injection site bruising (General disorders) | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 1 | 3 | 0
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 80 | 50 | 58 | 85
Injection site scar (General disorders) | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Polyp (General disorders) | 1 | 0 | 0 | 0
Pyrexia (FEVER) (General disorders) | 13 | 6 | 10 | 8
Swelling (SWELLING) (General disorders) | 20 | 2 | 1 | 13
Vaccination site pain (General disorders) | 3 | 0 | 3 | 0
Vessel puncture site bruise (General disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 5
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 57 | 32 | 43 | 43
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (NAUSEA) (Gastrointestinal disorders) | 53 | 32 | 42 | 37
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (VOMITING) (Gastrointestinal disorders) | 7 | 3 | 4 | 8
Allergy to vaccine (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Asymptomatic COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 5 | 0 | 3
COVID-19 (Infections and infestations) | 36 | 30 | 27 | 20
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Dacryocanaliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 2 | 2
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 2 | 2
Localised infection (Infections and infestations) | 1 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 2 | 3 | 0
Nasal herpes (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 4
Respiratory tract infection viral (Infections and infestations) | 1 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 3 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 16 | 13 | 23 | 15
Urinary tract infection (Infections and infestations) | 2 | 1 | 2 | 2
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 9 | 4 | 2 | 3
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Chemical burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 4 | 3 | 5
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Biopsy breast (Investigations) | 1 | 0 | 0 | 0
Biopsy skin (Investigations) | 0 | 0 | 0 | 1
Blood testosterone decreased (Investigations) | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 2
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 81 | 50 | 64 | 49
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 111 | 61 | 85 | 65
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anosmia (Nervous system disorders) | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 3 | 3 | 2
Headache (HEADACHE) (Nervous system disorders) | 138 | 103 | 145 | 111
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 2
Presyncope (Nervous system disorders) | 0 | 2 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Ulnar neuritis (Nervous system disorders) | 1 | 0 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast calcifications (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 21 | 3 | 5 | 11
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT05301322/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT05301322/SAP_001.pdf